CLINICAL TRIAL: NCT05899140
Title: Adjunctive Clindamycin Versus Standard of Care for the Treatment of Skin and Soft Tissue Infections, a Randomized Controlled, Open-label Superiority Phase 4 Trial
Brief Title: Adjunctive Clindamycin for the Treatment of Skin and Soft Tissue Infections, a Randomized Controlled Trial
Acronym: SoTiClin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Frieder Schaumburg (Other)
Responsible Party: Sponsor-Investigator, Frieder Schaumburg, Principal Investigator, Professor, Universität Münster
Organization: Universität Münster (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SoTiClin
Record Dates: First submitted 2023-05-22; First posted 2023-06-12 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Skin Infection; Staphylococcal Infections; Staphylococcus Aureus Infection
Keywords: SSTI; Staphylococcus aureus; Panton-Valentine leukocidin
MeSH Terms: conditions — Cellulitis; Staphylococcal Infections | interventions — Clindamycin; Standard of Care

STUDY DESIGN:
Intervention Model Description: 2-arm randomized controlled trial
Masking Description: This is an exploratory study and will not use a placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Other): Participants with skin and soft-tissue infections requiring systemic treatment (oral or intravenous). Treatment according to local guidelines = standard of care: usually an anti-staphylococcal penicillin with or without incision and drainage, as required.
  Treatment can be with (local guidelines) cloxacillin (non-severe) po 500g QIDfor 5-7 days ceftriaxone (severe infections) 2g iv OD with step-down to cloxacillin po 500 mg QID for a total of 7 days
  Interventions: Other: Standard of care
- Standard of care + clindamycin (Active Comparator): Participants with skin and soft-tissue infections requiring systemic treatment (oral or intravenous).
  Addition of clindamycin: 10 mg/kg/dose QID iv (maximum 600mg QID iv) or oral clindamycin 450 mg TDS for adults for a total of 7 days from randomisation.
  Interventions: Drug: Clindamycin; Other: Standard of care

INTERVENTIONS:
Drug: Clindamycin — Clindamycin will be administered at a dose of 450 mg TDS (oral) or 10 mg/kg/dose QID iv (maximum 600mg QID iv) for a maximum of 7 days
  Arms: Standard of care + clindamycin
Other: Standard of care — Standard of care

SUMMARY:
This is an exploratory study to evaluate the effect of adjunctive clindamycin in the treatment of skin and soft-tissue infections due to Staphylococcus aureus in patients from Sierra Leone. The study hypothesizes that clindamycin, when added to routine treatment, will lead to a more rapid clinical resolution and less frequent recurrences of infection.

DETAILED DESCRIPTION:
Panton-Valentine Leukokidin and other toxins play an important role in the severity of skin and soft-tissue infections due to Staphylococcus aureus. The inhibition of the protein synthesis could be beneficial, due to the major role of protein-toxins in the pathogenesis of skin and soft tissue infections. Clindamycin has a strong toxin-suppressive activity. Therefore, clindamycin is currently considered as the most-promising adjuvant antimicrobial agent in the treatment of toxin-mediated S. aureus infections. Recurrent infections are common in patients with S. aureus skin and soft-tissue infections. Clindamycin has been reported to reduce S. aureus colonisation, which may in turn reduce the risk for recurrent infections. Clindamycin is an already approved antimicrobial used for a wide range of indications and with a known safety profile.

This study is an investigator-led, investigator-initiated, open-label superiority randomised controlled trial that will be conducted at Masanga Hospital in Sierra Leone. The objectives of this study are to determine the feasibility, efficacy and safety of adjunctive clindamycin therapy (in addition to standard-of-care) compared to standard-of-care alone on clinical treatment outcomes in patients with skin and soft tissue infections due to S. aureus in Sierra Leone. This is a preliminary study, which will include 100 adult participants with skin and soft-tissue infections requiring systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥18 years);
2. Need for a treatment (incision/drainage ± antibiotic treatment po or iv) of an SSTI;
3. S. aureus causing SSTI identified from at least one clinical specimen (including isolation in polymicrobial cultures if S. aureus is considered to be the leading pathogen);
4. Onset of symptoms within the last 4 weeks;
5. Randomisation possible within 72 hours from collection of the initial culture
6. Ability to conduct the follow-up visits either during admission or at home
7. Initial culture collected within 48 hours of hospital admission
8. Willingness to participate in the study.

Exclusion Criteria

1. Previous allergic reaction to clindamycin
2. Previous antibiotic-associated diarrhea
3. Previous study participation
4. Pregnancy as confirmed by a beta-HCG rapid test.
5. Started treatment with clindamycin prior to clinic presentation;
6. Documented systemic antibiotic treatment within the previous 14 days
7. Co-administration of other protein synthesis inhibitors (e.g. macrolides, rifampicin, linezolid, aminoglycosides, tetracyclines, chloramphenicol);
8. Co-administration of toxin inducers (trimethoprim-sulfamethoxazole)
9. Severe illness (patient expected to die in the following 24 hrs);
10. Chronically infected wounds (>4 weeks of symptoms);
11. Infections associated with any of the following (due to mixed infection): a) Human or animal bites;b) Prosthetic or implantable devices; c) Decubitus ulcers; d) Diabetic foot ulcers, infected ulcers secondary to peripheral artery disease, chronic venous insufficiency; e) Suspected Buruli ulcer; f) Infected burns.
12. Hospital-acquired infection including post-surgical site infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical cure at follow-up 7 days | Day 7
  Proportion of patients with clinical cure defined as the absence of clinical failure

SECONDARY OUTCOMES:
Change in inflammatory markers under therapy | from baseline to Day 3 and from baseline to Day 7
  Change in mean C-reactive protein level
Time to symptom resolution | during follow-up up to day 14
  Time to resolution of symptoms
Occurence of adverse events | anytime during follow-up (to day 14)
  Proportion of patients with adverse events (of any kind) and of adverse events that required treatment discontinuation or change in drugs used
Microbiological failure | during follow-up day 3 and day 7
  Proportion of microbiological treatment failure (culture of S. aureus in relevant materials) on Day 3 and Day 7;
Clostridioides difficile associated diarrhoea | during follow-up, up to day 14
  Proportion with Clostridioides difficile associated diarrhoea
Recurrent infections | 6 months passive follow-up (participant re-presents to clinic)
  Proportion of recurrent infections during a passive follow up of 6 months
Clinical cure at follow-up 14 days | Day 14
  Proportion of patients with clinical cure defined as the absence of clinical failure

CONTACTS AND LOCATIONS:
Overall Officials: Frieder Schaumburg, MD, Principal Investigator — Universität Münster
Locations (1):
- Masanga Hospital, Masokori, Sierra Leone

IPD SHARING:
Plan to Share IPD: No
This is currently being considered and the information will be updated once a decision has been reached